CLINICAL TRIAL: NCT06043700
Title: A Community-Based Screening Program to Identify, Using Blood-Based Biomarkers, Individuals With or Without Alzheimer's Disease Symptoms Who Are at High Risk for Brain Amyloid Pathology
Brief Title: A Community-Based Screening Program to Identify Participants at High Risk for Amyloid Pathology
Status: Enrolling by invitation | Type: Observational
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: R2000-G000-008
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimers Disease; Blood-based biomarkers; Community-based screening
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual blood samples will be retained after obtaining consent from the participants and may be used for future biomarker assessment for AD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants with or without symptoms of AD will be enrolled and observed in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No treatment intervention will be administered.

SUMMARY:
The primary purpose of this study is to identify participants with or without symptoms of Alzheimer's Disease (AD) that are at high risk for brain amyloid pathology using blood-based biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 50 to 80 years inclusive, at the time of informed consent

   - Those 50 to 64 years of age must have 1 of the following risk factors confirmed prior to blood sample collection:
   * First degree relative with dementia onset before age 75,
   * Known before screening to have at least 1 Apolipoprotein E4 (APOE4) allele, or
   * Known before screening to have elevated brain amyloid according to previous positron emission tomography (PET), cerebrospinal fluid (CSF), or blood testing
2. Provide written informed consent
3. Willing and able to comply with all aspects of the protocol
4. Willing to be referred to a clinical site if the assessment results meet the criteria

Exclusion Criteria:

1. Known uncontrolled medical conditions (example, cardiac, respiratory, gastrointestinal, psychiatric, renal disease, malignant neoplasm)
2. Participation in an interventional clinical trial study at the time of consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with or without symptoms of AD will be screened in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Low, Medium, and High Amyloid Pathology | At Screening on Day 1
  Number of participants with low, medium, and high amyloid pathology will be estimated.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Eisai Site #3, Clermont, Florida
  - Eisai Site #1, Lady Lake, Florida
  - Eisai Site #2, District Heights, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.